CLINICAL TRIAL: NCT03256110
Title: Exploring Palliative Care Communication With Alaska Native and American Indian People at Two Sites
Brief Title: Palliative Care Communication With Alaska Native and American Indian People
Acronym: PALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southcentral Foundation (Other)
Collaborators: University of Colorado, Denver (Other); University of New Mexico (Other); Washington State University (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Jennifer Shaw, Senior Researcher, Southcentral Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R21NR016611 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Advance Care Planning
Keywords: Advance Care Planning; Palliative Care; Indians, North American; Alaska Natives; Health Communication; Primary Health Care

STUDY DESIGN:
Intervention Model Description: Cluster-randomized design with providers randomized to intervention or control and patients nested within provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients and providers in this arm receive the culturally-tailored Improving Communication about Serious Illness (ICSI) Intervention. The ICSI involves providing the provider and the patient with an individualized, one-page summary of patient-specific preferences for advance care planning communication that prompts the patient and the provider to have a conversation about advance care planning at the next clinical visit.
  Interventions: Behavioral: Improving Communication about Serious Illness-AI/AN
- Control (No Intervention): Patients and providers in this arm receive usual care.

INTERVENTIONS:
Behavioral: Improving Communication about Serious Illness-AI/AN — A one-page summary of patient-specific preferences, barriers and facilitators for engaging in patient-provider communication about advance care planning, provided to patient and provider prior to a clinical encounter with prompts for initiating and/or improving the quality of communication about advance care planning.
  Arms: Intervention

SUMMARY:
This mixed-methods study is culturally tailoring and evaluating a communication intervention to increase the frequency and quality of advance care planning with diverse American Indian and Alaska Native adults with serious, life-limiting illness in primary care at two sites.

DETAILED DESCRIPTION:
Palliative care is an interdisciplinary field that aims to relieve emotional, spiritual and physical suffering and improve quality of life in patients with serious, life-limiting illness and their families. Unfortunately, palliative care is often introduced too late in the course of care to maximize its potential benefits, in part because healthcare providers and patients alike lack the knowledge and self-efficacy to initiate conversations about advance care planning (ACP). ACP is an important component of palliative care in which patients, families and providers discuss and plan for the patient's desired treatment goals, including preferences for care and who can make decisions on the patient's behalf if needed. Integrating ACP into treatment early, before serious, life-limiting illness advances to a late stage, can improve patient and caregiver quality of life, length of survival, and health care cost. Primary care is an ideal setting for early integration of ACP, as primary care providers routinely diagnose and care for patients in the early stage of serious, life-limiting conditions, such as chronic obstructive pulmonary disease. Alaska Native and American Indian (AN/AI) people have disproportionately high prevalence of many serious, life-limiting conditions, including cancer, coronary heart disease, and liver disease. Yet, AN/AIs use ACP and other palliative care services significantly less than the overall population. The reasons for this disparity are unclear, and AN/AIs are among the most underrepresented groups in palliative care studies. Previous research indicates that when given the opportunity, AIs will engage in ACP, and our preliminary data suggest strong support among ANs for developing culturally congruent ACP interventions in primary care settings. The need for timely and effective ACP is growing in AN/AI communities and there is a pressing need for culturally-congruent, patient-centered palliative care interventions for AN/AIs as tribal health systems manage rising numbers of AN/AI individuals with serious, life-limiting illnesses. The aims of this collaborative, community-engaged, clinical study are to: 1) conduct focus groups with 40 key stakeholders (patients, caregivers, providers, administrators) in two tribal health systems to tailor an existing ACP communication intervention for AN/AIs with serious, life-limiting illness; 2) evaluate the cultural relevance and usability of the tailored ACP communication intervention among 20 AN/AI patients using cognitive interviews; and 3) compare the impact of the tailored intervention on frequency of ACP discussions, as well as quality of and satisfaction with ACP communication between 30 AN/AI patients receiving individualized information to prompt ACP discussions with providers and 30 AN/AI patients receiving usual care, with information to prompt a discussion. Implementing effective, appropriate ACP is a high priority at Southcentral Foundation (SCF) and First Nations Community HealthSource (FNCH), two tribal health systems serving large, diverse populations of AN/AI people in Alaska and New Mexico. This study will develop and evaluate a culturally congruent, patient- centered ACP intervention at these sites and produce evidence for a large, multi-site clinical trial of the intervention that could improve patient and caregiver outcomes in this diverse population of more than 5 million Americans.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native and/or American Indian (patients)
* Age 18 or older (patients and providers)
* Employed at least 2 years as a primary care provider at one of the two study sites (providers)
* Have a primary care provider of record at one of the two study sites (patients)
* Have had at least 2 visits with primary care provider in previous 12 months (patients)
* Having at least one serious, life-limiting condition, including metastatic cancer, primary lung cancer, chronic obstructive pulmonary disorder, heart disease, liver disease or cirrhosis, renal failure, or being oxygen dependent. (patients)

Exclusion Criteria:

* Under age 18 (patients and providers)
* Not Alaska Native or American Indian (patients)
* Not having a primary care provider at one of the study sites (patients)
* Not being employed for at least two years as a primary care provider at one of the study sites (providers)
* Not having had at least 2 visits with a primary care providers at one of the study sites in the previous 12 months (patients)
* Not having a serious, life-limiting condition, such as metastatic cancer, primary lung cancer, chronic obstructive pulmonary disorder, heart disease, liver disease or cirrhosis, renal failure, or being oxygen dependent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
ACP communication occurrence | up to 2 weeks
  Patient self-report of occurence of advance care planning communication.
ACP communication quality | up to 2 weeks
  Patient self-report of quality of advance care planning communication

SECONDARY OUTCOMES:
Advance Directives | up to 1 month
  Documentation of advance directives (i.e. health care agent and living will) in electronic health record

OTHER OUTCOMES:
Intervention feasibility-provider | up to 1 week
  Provider self-report of ease of using advance care planning communication tool
Intervention feasibility-patient | up to 2 weeks
  Patient self-report of ease of using advance care planning communication tool
Intervention acceptability-provider | up to 1 week
  Provider self-report of cultural acceptability of advance care planning communication tool
Intervention acceptability-patient | up to 2 weeks
  Patient self-report of cultural acceptability of advance care planning communication tool

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Shaw, PhD, Principal Investigator — Southcentral Foundation
Locations (2):
- United States (2):
  - Southcentral Foundation, Anchorage, Alaska
  - First Nations Community HealthSource, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No